CLINICAL TRIAL: NCT04010617
Title: Pharyngeal Electrical Stimulation (PES) to Avoid Extubation Failure in Intubated Stroke at High Risk of Severe Dysphagia
Brief Title: PES to Avoid Extubation Failure in Intubated Stroke Patients at High Risk of Severe Dysphagia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01072018
Record Dates: First submitted 2019-05-29; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-05

CONDITIONS: Stroke; Dysphagia; Extubation Failure
Keywords: Pharyngeal Electrical Stimulation; Stroke; Dysphagia; Re-intubation
MeSH Terms: conditions — Stroke; Deglutition Disorders

STUDY DESIGN:
Intervention Model Description: Observational trial with comparison to a historical control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharyngeal Electrical Stimulation (Experimental): Orotracheal intubated patients at high risk of extubation failure will receive open-label PES
  Interventions: Device: Pharyngeal Electrical Stimulation (PES)

INTERVENTIONS:
Device: Pharyngeal Electrical Stimulation (PES) — PES will be delivered by a commercial device (Phagenyx, Phagenesis Ltd, Manchester, UK), which comprises a nasogastric feeding catheter that houses stimulation ring-electrodes and a computerised base station that delivers stimulation in the range 1-50 mA at 5 Hz.

SUMMARY:
Post-extubation dysphagia (PED) recently became a growing concern as a major risk factor for extubation failure and significant contributor to poor patient outcomes with prevalence rates ranging from 12% to 69%, being highest in neurological patients (93%).

Pharyngeal electrical stimulation (PES) has been shown to improve airway safety and swallowing function tracheostomized stroke patients, thereby enhancing decannulation in this patient cohort.

In the present study the investigators evaluate whether PES is safe, feasible and effective in orotracheal intubated stroke patients at high risk of extubation failure.

DETAILED DESCRIPTION:
Endotracheal intubation and mechanical ventilation are common procedures for critically ill stroke patients. Although necessary and life-saving, timely extubation after ventilator weaning is desirable, because patients with delayed extubation experience higher pneumonia rate, increased need for tracheostomy, longer length of stay on the intensive care unit and higher mortality. On the other hand, extubation failure (EF) and subsequent need for emergent re-intubation is associated with similar sequelae.

Post-extubation dysphagia (PED) became a growing concern as a major risk factor for EF and significant contributor to poor patient outcomes with prevalence rates ranging from 12% to 69%, being highest in neurological patients (93%). Damage to the central swallowing network itself is the primary cause of PED in cerebrovascular disease, which constitutes the leading diagnosis on neuro-ICUs. Further mechanisms include pharyngolaryngeal lesions caused by the tube, critical illness neuropathy and myopathy leading to muscle weakness and dyscoordination of breathing and swallowing, and an impaired sensation due to sedation, mucosal damage, or the underlying critical illness itself. As a consequence reintubation rates in neurological collectives are as high as 20 to 40%.

Pharyngeal electrical stimulation (PES) has been shown to improve airway safety and swallowing function tracheostomized stroke patients, thereby enhancing decannulation in this patient cohort.

In the present study the investigators evaluate whether PES is safe, feasible and effective in orotracheal intubated stroke patients at high risk of extubation failure.

ELIGIBILITY:
Inclusion Criteria:

Acute stroke orotracheal intubation high-risk of extubation failure (DEFISS-score ≥4) successful respiratory weaning according to the treating intensivist within 24 to 72 hours

Exclusion Criteria:

Patients are excluded from study participation if any of the following apply:

* Suffer from pre-existing neurogenic dysphagia or a condition that can cause dysphagia (for example Parkinson's Disease);
* Suffer from non-neurogenic dysphagia (e.g. cancer);
* Suffer from neuromuscular disorders (e.g. myasthenia gravis, motor neuron disease);
* Participate in any other study potentially influencing the outcome of PES, both medicinal or medical device product related and for which the patient signed a consent form for his/her study participation;
* Receive or have received within one month prior to the intended PES treatment any other type of standard cranial or percutaneous electrical stimulation therapy to treat dysphagia;
* Have a pacemaker or an implantable defibrillator;
* Have a nasal anatomical deformity, nasal airway obstruction, have had oesophageal surgery or any other circumstance where placement of a standard NG feeding tube would be deemed unsafe;
* Have a cardiac or respiratory condition that might render the insertion of the catheter into the throat unsafe;
* Are pregnant or nursing women;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Successful extubation | 72 hours after extubation
  No re-intubation within 72 hours after extubation

SECONDARY OUTCOMES:
Pneumonia | up to 14 days
  Pneumonia post extubation until hospital discharge
Feeding status | up to 14 days
  Functional Oral Intake Scale
Swallowing function | 0-24 hours after extubation
  Fiberoptic Endoscopic Dysphagia Severity Scale
Swallowing function | 72-120 hours after extubation
  Fiberoptic Endoscopic Dysphagia Severity Scale
Swallowing function | up to 14 days
  Fiberoptic Endoscopic Dysphagia Severity Scale
Length of stay of the ICU/intermediate care | up to 60 days
  Length of stay in days
Length of stay in hospital | up to 120 days
  Length of stay in hospital in days

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Dziewas, MD, Principal Investigator — Department of Neurology, University Hospital Münster, Germany
Locations (1):
- University Hospital Münster, Deparment of Neurology, Münster, Germany

IPD SHARING:
Plan to Share IPD: No
a subset of fully anonymised patient data may be available upon request from the authors